CLINICAL TRIAL: NCT02931461
Title: Interest of Procore Needle® for Diagnosis of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR-EBUS
Record Dates: First submitted 2016-09-07; First posted 2016-10-13 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Endobronchial Transbronchial Needle Aspiration Lung Cancer Procore
Keywords: endobronchial transbronchial needle aspiration lung cancer procore

ARMS (2):
- needle Procore ® (Experimental)
  Interventions: Procedure: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration
- needle Cook® (Active Comparator)
  Interventions: Procedure: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration

INTERVENTIONS:
Procedure: Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration

SUMMARY:
The ProCore ultrasound biopsy needle, used primarily to obtain intra-abdominal tissue core biopsies, has not been widely used for endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA). In this study the investigators are going to evaluate the utility of the ProCore needle for sampling mediastinal or hilar lymph nodes during EBUS-TBNA versus standard 22 gauge needle for diagnosis of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* mediastinal lymphadenopathy >10 millimeters
* lung cancer suspected

Exclusion Criteria:

* coagulopathy contraindication for midazolam contraindication for bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Proportion of histological diagnoses for each needle | 6 months